CLINICAL TRIAL: NCT01079728
Title: Prediction of Stroke-associated Pneumonia
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Siemens Health Care (Unknown); NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Professor Dr. med., Charite University, Berlin, Germany
Other Study IDs: PREDICT
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; stroke-associated pneumonia; prediction; immune and infection parameters
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample (serum, plasma)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ischemic stroke patients: patients with an ischemic stroke in the anterior (ACA, MCA) and posterior flow area (PCA, BA) of any severity in the last 36h

SUMMARY:
Stroke-associated pneumonia (SAP) constitutes a clinically relevant complication of stroke, because it increases the mortality and has a negative impact on the neurological prognosis of the patient.

An early identification of patients at risk for SAP allowing an early initiation of antiinfective therapy may improve the prognosis. To date, no reliable prediction models or clinical scores for stroke-associated pneumonia exist. Recently, it was shown that parameters indicating an impaired immune function are associated with the subsequent occurrence of SAP and could therefore be used as predictors for SAP.

This study will develop and prospectively validate a prognostic score to predict SAP based on clinical parameters. Furthermore, the study examines the prognostic properties of selected immune and infectious parameters for the prediction and diagnosis of SAP. The study will further address the question whether these infectious and immune parameters predict the 3-month-outcome. In a subgroup of patients, MRI parameters on stroke size and localization will be assessed to investigate whether these parameters might allow prediction of SAP or the 3-month-outcome.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke in the anterior (ACA, MCA) and posterior cerebral circulation (PCA, BA) of any severity
* stroke onset within the last 36h
* age ≥ 18
* consent by the patient or the legal representative

Exclusion Criteria:

* intracranial hemorrhage
* signs of infection at admission (clinical / paraclinical)
* pre-existing dysphagia
* mechanical ventilation at admission
* participation in an interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ischemic stroke in the anterior (ACA, MCA) and posterior cerebral circulation (PCA, BA) of any severity in the last 36h
Sampling Method: Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Predictive score for SAP based on clinical parameters assessed within 36h after stroke onset | SAP within 7 days after onset of symptoms (stroke)
  To establish a predictive score for SAP based on clinical parameters assessed within 36h after stroke onset
Predictive properties of immune parameters (IL6, IL10, mHLA-DR) or infection parameters (PCT) for the occurrence of a SAP within 7 days after stroke onset | SAP within 7 days after onset of symptoms (stroke)
  To evaluate of the predictive properties of immune parameters (IL6, IL10, mHLA-DR) or infection parameters (PCT) for the occurrence of a SAP within 7 days after stroke onset

SECONDARY OUTCOMES:
Predictive properties of immune parameters (IL6, IL8, IL10, mHLA-DR, MBL, monocytic cytokine secretion after ex vivo stimulation, C5a) and infection parameters (PCT, LBP) for the neurological outcome | Neurological outcome 3 months after onset of symptoms (stroke)
  To evaluate of the predictive properties of immune parameters (IL6, IL8, IL10, mHLA-DR, MBL, monocytic cytokine secretion after ex vivo stimulation, C5a) and infection parameters (PCT, LBP) for the neurological outcome
Plasma levels of acetylcholinesterase | within 7 days after onset of symptoms (stroke)
  To investigate the parasympathetic influence on the immune function after stroke by measuring plasma levels of acetylcholinesterase
Localization and stroke volume analysis | SAP within 7 days and neurological outcome after 3 months after onset of symptoms (stroke)
  To investigate the influence of the localization and stroke volume on the occurrence of a SAP and on neurological outcome
Predictive properties of immune parameters (IL6, IL8, IL10, mHLA-DR, MBL, monocytic cytokine secretion after ex vivo stimulation, C5a) and infection parameters (PCT, LBP) for the occurence of a SAP | SAP within 7 days after onset of symptoms (stroke)
  To evaluate of the predictive properties of immune parameters (IL6, IL8, IL10, mHLA-DR, MBL, monocytic cytokine secretion after ex vivo stimulation, C5a) and infection parameters (PCT, LBP) for the occurence of a SAP
Influence of insular cortex involvement and infarct volume on the occurrence of a SAP within 7 days and and on the neurological outcome after 3 months | SAP within 7 days after onset of symptoms (stroke) and neurological outcome after 3 months
  To investigate the influence of insular cortex involvement and infarct volume on the occurrence of a SAP within 7 days after stroke onset and on the neurological outcome after 3 months
Transcriptome analyses | SAP within 7 days and neurological outcome after 3 months after onset of symptoms (stroke)
  To perform transcriptome analyses to identify new biomarkers which may predict the occurence of a SAP or the 3-month neurological outcome

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, MD, Principal Investigator — Charite University Berlin (Center for Stroke Research Berlin CSB & NeuroCure Clinical Research Center NCRC); Peter Heuschmann, MD, Principal Investigator — Charité University Berlin (Center for Stroke Research Berlin CSB)
Locations (8):
- Germany (7):
  - Charite University (Center for Stroke Research Berlin CSB & NeuroCure Clinical Research Center NCRC), Berlin
  - Unfallkrankenhaus Berlin, Neurologie, Berlin
  - Vivantes Auguste Viktoria Klinikum Neurologie, Berlin
  - Vivantes Klinikum im Friedrichshain Neurologie, Berlin
  - Vivantes Klinikum Spandau Neurologie, Berlin
  - Vivantes Neukölln Neurologie, Berlin
  - Sankt Josefs Krankenhaus Potsdam Neurologie, Potsdam
- Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Hoffmann S, Harms H, Ulm L, Nabavi DG, Mackert BM, Schmehl I, Jungehulsing GJ, Montaner J, Bustamante A, Hermans M, Hamilton F, Gohler J, Malzahn U, Malsch C, Heuschmann PU, Meisel C, Meisel A; PREDICT Investigators. Stroke-induced immunodepression and dysphagia independently predict stroke-associated pneumonia - The PREDICT study. J Cereb Blood Flow Metab. 2017 Dec;37(12):3671-3682. doi: 10.1177/0271678X16671964. Epub 2016 Oct 14. PMID 27733675
- [Result] Hotter B, Hoffmann S, Ulm L, Meisel C, Bustamante A, Montaner J, Katan M, Smith CJ, Meisel A. External Validation of Five Scores to Predict Stroke-Associated Pneumonia and the Role of Selected Blood Biomarkers. Stroke. 2021 Jan;52(1):325-330. doi: 10.1161/STROKEAHA.120.031884. Epub 2020 Dec 7. PMID 33280547
- [Result] Hotter B, Hoffmann S, Ulm L, Meisel C, Fiebach JB, Meisel A. IL-6 Plasma Levels Correlate With Cerebral Perfusion Deficits and Infarct Sizes in Stroke Patients Without Associated Infections. Front Neurol. 2019 Feb 15;10:83. doi: 10.3389/fneur.2019.00083. eCollection 2019. PMID 30828313
- [Result] Hotter B, Hoffmann S, Ulm L, Montaner J, Bustamante A, Meisel C, Meisel A. Inflammatory and stress markers predicting pneumonia, outcome, and etiology in patients with stroke: Biomarkers for predicting pneumonia, functional outcome, and death after stroke. Neurol Neuroimmunol Neuroinflamm. 2020 Feb 25;7(3):e692. doi: 10.1212/NXI.0000000000000692. Print 2020 May. PMID 32098866
- [Result] Mengel A, Ulm L, Hotter B, Harms H, Piper SK, Grittner U, Montaner J, Meisel C, Meisel A, Hoffmann S. Biomarkers of immune capacity, infection and inflammation are associated with poor outcome and mortality after stroke - the PREDICT study. BMC Neurol. 2019 Jul 3;19(1):148. doi: 10.1186/s12883-019-1375-6. PMID 31269910
- [Result] Winek K, Lobentanzer S, Nadorp B, Dubnov S, Dames C, Jagdmann S, Moshitzky G, Hotter B, Meisel C, Greenberg DS, Shifman S, Klein J, Shenhar-Tsarfaty S, Meisel A, Soreq H. Transfer RNA fragments replace microRNA regulators of the cholinergic poststroke immune blockade. Proc Natl Acad Sci U S A. 2020 Dec 22;117(51):32606-32616. doi: 10.1073/pnas.2013542117. Epub 2020 Dec 7. PMID 33288717